CLINICAL TRIAL: NCT02796183
Title: The Efficacy of Subconjunctival Bevacizumab in Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neon Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Volkan YETER, MD, Neon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetic macular edema (Other): Bevacizumab (Altuzan) was injected subconjunctival space of the patients.
  Interventions: Drug: Subconjunctival bevacizumab (Altuzan)

INTERVENTIONS:
Drug: Subconjunctival bevacizumab (Altuzan) — Subconjunctival injections of Altuzan 3.75mg were applied in order to eliminate the macular edema.

SUMMARY:
This study evaluates the effects of subconjunctivally injected bevacizumab in patients with diffuse diabetic macular edema.

DETAILED DESCRIPTION:
At baseline, the macular thicknesses of both eyes of the patients with persistant diabetic macular edema were measured by optical coherence tomography. After 3.75mg bevacizumab was injected into subconjunctival space of the eyes with diabetic macular edema. The measurements of the macular thicknesses were repeated by optical coherence tomography in 15th, 30th, 60th day after injections. The macular thickness measurements before and after injection were compared.

ELIGIBILITY:
Inclusion Criteria:

* Having diffuse diabetic macular edema persisted at least 1 month
* No intravitreal injection in last 3 months.
* No retinal laser photocoagulation in last 6 months
* Not have any other macular disease causing macular edema

Exclusion Criteria:

* Having ischemic macula
* Intravitreal injection in last 3 months.
* Retinal laser photocoagulation in last 6 months
* Have any other macular disease causing macular edema

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Central Macular Thickness | one year (between May 2015 and May 2016)

IPD SHARING:
Plan to Share IPD: No